CLINICAL TRIAL: NCT02940821
Title: Assessing Three Oral Care Regimen on Plaque, Gingivitis, and Tooth Whitening
Brief Title: Assessing the Effects of Three Oral Care Regimens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pearl Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PRL1517
Record Dates: First submitted 2016-10-06; First posted 2016-10-21 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Dental Plaque; Gingivitis
Keywords: Tooth Whitening
MeSH Terms: conditions — Dental Plaque; Gingivitis | interventions — Toothbrushing; fluorophosphate; Tin Fluorides; Hydrogen Peroxide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Whitening and Dentifrice (Active Comparator)
  Interventions: Other: Toothbrushing; Other: Whitening (4.5% hydrogen peroxide); Other: Other Fluoridated Dentifrice (.454% stannous fluoride)
- Whitening Dentifrice (Active Comparator)
  Interventions: Other: Toothbrushing; Other: Fluoridated Dentifrice Whitening System (.454% stannous fluoride with 2% hydrogen peroxide)
- Dentifrice (Active Comparator)
  Interventions: Other: Toothbrushing; Other: Fluoridated Dentifrice (.15% sodium monofluorophosphate)

INTERVENTIONS:
Other: Toothbrushing — Mechanical plaque removal
  Other Names: Toothbrush
Other: Fluoridated Dentifrice (.15% sodium monofluorophosphate) — Fluoridated dentifrice application
  Arms: Dentifrice
Other: Fluoridated Dentifrice Whitening System (.454% stannous fluoride with 2% hydrogen peroxide) — Application of Tooth Whitening Agent in Dentifrice
  Other Names: Fluoridated Dentifrice Whitening System (.454% stannous fluoride with 2% hydrogen peroxide) and toothbrushing
  Arms: Whitening Dentifrice
Other: Whitening (4.5% hydrogen peroxide) — Application of Whitening Agent
  Arms: Whitening and Dentifrice
Other: Other Fluoridated Dentifrice (.454% stannous fluoride) — Fluoridated dentifrice application
  Other Names: Fluoridated dentifrice (.454% stannous fluoride)
  Arms: Whitening and Dentifrice

SUMMARY:
Assessing the effects of three oral care regimen on plaque, gingivitis, and tooth whitening: A randomized, person-centric, comparative effectiveness clinical research study by the Practitioners Engaged in Applied Research and Learning (PEARL) Network.

DETAILED DESCRIPTION:
Six month, five visit study of plaque, gingivitis, and tooth whitening with three randomized intervention groups using FDA marketed and approved products and devices. One hundred fifty (150) subjects from the patient base of 10 PEARL Network associated dental offices on the East Coast of the United States will be entered into the clinical research study. This is a post-marketing comparative effectiveness research study. Having a total of 5 visits over a six month period. Adverse events and side effects for the products used are being assessed.

ELIGIBILITY:
Inclusion Criteria

1. Subject males or females 18 to 70 years old (inclusive).
2. Availability for the 6 months duration of the clinical research study
3. Good general health
4. Subject able and willing to follow study procedures and instructions
5. Subject read, understood and signed an informed consent form
6. Subject present with at least 20 natural teeth in the functional dentition (excluding third molars), including the following natural (uncrowned) teeth for shading: #6, #7, #8, #9, #10, #11

Exclusion Criteria

Potential subjects must NOT HAVE ANY of the following conditions:

1. Presence of orthodontic bands
2. Presence of partial removable dentures
3. Tumor(s) of the soft or hard tissues of the oral cavity
4. Restorations or crowns that would interfere with color measurements on the following teeth: #6, #7, #8 , #9, #10 & #11 (upper six front teeth)
5. Advanced periodontal disease (purulent exudate, tooth mobility, and/or extensive loss of periodontal attachment or alveolar bone)
6. Five or more carious lesions requiring immediate restorative treatment
7. Antibiotic use any time during the one month prior to entry into the study
8. Participation in any other clinical study or test panel within the one month prior to entry into the study
9. History of allergies to oral care/personal care consumer products or their ingredients.
10. On any prescription medicines that might interfere with the study outcome
11. An existing medical condition which prohibits eating or drinking for periods up to 4 hours
12. History of alcohol or drug abuse
13. Pregnant or lactating

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2016-05-30 (Actual); Primary Completion 2017-07-27 (Actual); Study Completion 2017-07-27 (Actual)

PRIMARY OUTCOMES:
Tooth Whitening Shade Evaluation | 6 months

SECONDARY OUTCOMES:
Patient Questionnaire | 6 months
Plaque Index | 6 months
Gingival Index | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Frederick A Curro, DMD, PhD, Study Director — Pearl Network; Ashley C Grill, MPH, RDH, Principal Investigator — Pearl Network
Locations (1):
- Frederick A. Curro, DMD, PhD, Emerson, New Jersey, United States